CLINICAL TRIAL: NCT04953117
Title: Assess the Safety and Efficacy of Lepu® Drug Coated Balloon Versus RESTORE® Paclitaxel Eluting Balloon for the Treatment of Coronary Small-vessel Disease: a Prospective, Multicenter, Randomized, Controlled Trial
Brief Title: A Safety and Efficacy Study of Lepu® Drug Coated Balloon in Treatment of Coronary Small-vessel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LP-SDCB-2020
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease
Keywords: Drug Coated Balloon Catheter; Small Coronary Vessel Disease; Randomized Controlled Trial
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- small vessel cohort: DCB of Lepu Medical (Experimental): receiving the treatment with DCB of Lepu Medical(dimeter≥2.00 mm) in small vessel cohort
  Interventions: Device: DCB of Lepu Medical(dimeter≥2.00 mm)
- small vessel cohort:Restore DEB (Active Comparator): receiving the treatment with Restore DEB in small vessel cohort
  Interventions: Device: Restore DEB
- very small vessel cohort: DCB of Lepu Medical (Other): receiving the treatment with DCB of Lepu Medical(dimeter<2.00 mm) in very small vessel cohort
  Interventions: Device: DCB of Lepu Medical(dimeter<2.00 mm)

INTERVENTIONS:
Device: DCB of Lepu Medical(dimeter≥2.00 mm) — subjects receiving DCB of Lepu Medical(dimeter≥2.00 mm)
  Other Names: Coronary Drug Coated Balloon Catheter of Lepu Medical for coronary small vessels
  Arms: small vessel cohort: DCB of Lepu Medical
Device: Restore DEB — subjects receiving Restore DEB
  Other Names: RESTORE Paclitaxel releasing coronary balloon catheter
  Arms: small vessel cohort:Restore DEB
Device: DCB of Lepu Medical(dimeter<2.00 mm) — subjects receiving DCB of Lepu Medical(dimeter<2.00 mm)
  Other Names: Coronary Drug Coated Balloon Catheter of Lepu Medical for coronary very small vessels
  Arms: very small vessel cohort: DCB of Lepu Medical

SUMMARY:
This study was designed to verify the safety and efficacy of Lepu® Drug Coated Balloon in Treatment of Coronary Small-vessel Disease

DETAILED DESCRIPTION:
This study include a small vessel cohort and a very small vessel cohort. In the small vessel cohort, patients with visually estimated reference vessel diameters(RVDs)≥2.0 and ≤2.75mm were randomly assigned to the Coronary Drug Coated Balloon Catheter Used in Small Vessels of Lepu Medical or the Restore DEB in a 1:1 ratio. The study was powered to detect the noninferiority of the DCB of Lepu Medical versus the Restore DEB for a primary endpoint of in-segment late lumen loss(LLL) at 9 months.

In the very small vessel cohort, patients with RVD≥1.75 and<2.0mm were treated with the DCB of Lepu Medical of an appropriate size.

All subjects will been followed up for 2 years to observe the occurrence of adverse events, so as to make an accurate and reliable evaluation of the safety of drug coated balloon catheters for coronary small vessels.

ELIGIBILITY:
Inclusion Criteria:

* Age must be 18-80 years, males or females.
* Subject with stable angina, or unstable angina, or recent myocardial infarction (myocardial infarction occurred more than 7 days before enrolled into the group), or asymptomatic myocardial ischemia with evidence
* Coronary angiopathy in situ with stenosis of more than 70% with visually estimated (or more than 50% combined with symptoms of ischemia, TIMI ≥ 1) in a vessel with visually estimated reference vessel diameter (RVD) ≥ 2.0 mm and ≤ 2.75 mm in small vessel group,and ≤ 26 mm in length or RVD ≥ 1.75 mm and < 2.0 mm in very small vessel group, and ≤ 16 mm in length.
* Target small vessel lesions are located on one or two different coronary arteries (RCA / LAD/ LCX). The number of target small vessel lesions on each coronary artery is no more than one, and each target small vessel lesion can only be treated with one test instrument
* The number of non-target lesions requiring early interventional treatment is no more than two, and the distance between them and target lesions must be > 10 mm; Successful treatment of non target lesions is required before subjects are randomized and the test equipment(DCB) cannot be used for the treatment.
* Subject can receive any type of coronary revascularization (including balloon angioplasty, stent implantation or coronary artery bypass grafting)
* Subject can understand the study objectives and voluntarily participate in and sign the informed consent; subject must agree to clinical follow-up and angiographic follow-up at 9 months.

Exclusion Criteria:

* AMI within 1 week.
* In stent restenosis, complete occlusion or severe calcification (unable to pre expand successfully with balloon)
* Left main artery disease or bifurcation disease with diameter >2.00mm requiring interventional treatment
* Evidence of massive thrombi in the target vessels
* Severe heart failure (NYHA IV)
* Severe renal failure (subject with GFR < 30ml / min or undergoing hemodialysis)
* Subject with vein graft restenosis after bypass surgery or severe heart valve disease
* Pregnant or nursing subjects
* Life expectancy less than 12 months
* Subject with bleeding tendency, history of active peptic ulcer, suffered stroke within the past 6 months, contraindications of antiplatelet preparation and anticoagulant treatment
* Subject is currently participating in another investigational drug or device study that has not yet completed its primary endpoint.
* Subject has undergone heart transplantation
* Known allergy to aspirin, clopidogrel, heparin, contrast media, and paclitaxel.
* The investigator judged that the subject's compliance is poor and can not complete the study as required.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
In-segment late lumen loss(LLL) | 9 months
  In-segment late lumen loss is defined as the change in minimal lumen diameter

SECONDARY OUTCOMES:
The success rate of intervention treatment (%)(Device success,Lesion success ,Procedural success) | 2-3 days
  The success rate of intervention treatment (%) include device success,lesion success and procedural success
In-segment diameter stenosis(DS%) | 9 months
  In-segment diameter stenosis(DS%) defined as (1-minimal luminal diameter[MLD]/reference vessel diameter[RVD])*100%.
Angiographic binary restenosis (ABR) | 9 months
  Angiographic binary restenosis (ABR), defined as target lesion DS ≥ 50% at follow up
Target lesion failure (TLF) | 30 days,6,9 months,and 1,2 years
  Target lesion failure (TLF), including cardiac death, target vessel-myocardial infarction (MI), or ischemic-driven target lesion revascularization (ID-TLR)
Patient-oriented composite endpoint (PoCE) | 30 days,6,9 months,and 1,2 years
  Patient-oriented composite endpoint (PoCE), including all-cause death, all MI, or any revascularization.
Definite or probable target lesion thrombosis | 30 days,6,9 months,and 1,2 years
  Definite or probable target lesion thrombosis, including Acute stent thrombosis, Early stent thrombosis, Late stent thrombosis, Very late stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Yida Tang, Study Chair — Peking University Third Hospital
Locations (14):
- China (14):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chao-Yang Hospital, Cpaital Medical University, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - No.980 Hospital of Joint Logistics Support Force, Shijiazhuang, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Inner Mongolia People's Hospital, Hohhot, Neimenggu
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital,School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang